CLINICAL TRIAL: NCT04868019
Title: Fenofibrate in Indirect Neonatal Hyperbilirubinemia
Brief Title: Role of Fenofibrate in Indirect Neonatal Hyperbilirubinemia: a Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Dr Nighat Haider, Assistant Professor, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.F.1-1/2015/ERB/SZABMU/654
Record Dates: First submitted 2021-04-29; First posted 2021-04-30 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Hyperbilirubinemia, Neonatal
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal | interventions — Fenofibrate

STUDY DESIGN:
Intervention Model Description: Groups A will receive Solution A i.e. Fenofibrate suspension is prepared by dissolving 200 mg capsule in 10 ml distilled water and given as a single dose of 10mg/kg (0.5 ml/kg) and Group B will receive solution B i.e. 0.5ml/ kg normal saline as a placebo. Both groups will receive LED phototherapy under standard conditions. The serum bilirubin level will be noted at the time of admission and then at 12hr, 24hr, and 48 hours of treatment.
Who Masked: Participant
Masking Description: Complete history and examination will be carried out while patients will be screened for enrollment. After taking informed consent, eligible patients will be selected and divided into two groups A and B by lottery method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Groups A will receive solution A .i.e fenofibrate suspension
  Interventions: Drug: Fenofibrate Capsules
- Group B (Placebo Comparator): Group B will receive solution B i.e placebo.
  Interventions: Drug: Fenofibrate Capsules

INTERVENTIONS:
Drug: Fenofibrate Capsules — Solutions will be prepared in the required strengths and labeled accordingly. Group A will receive Solution A i.e. Fenofibrate suspension is prepared by dissolving 200 mg capsule in 10 ml distilled water and given as a single dose of 10mg/kg (0.5 ml/kg) and Group B will receive solution B i.e. 0.5ml/ kg normal saline as a placebo. Both groups will receive LED phototherapy under standard conditions. The serum bilirubin level will be noted at the time of admission and then at 12hr, 24hr, and 48 hours of treatment
  Other Names: capsule fenoget

SUMMARY:
Fenofibrate accelerates bilirubin conjugation and excretion, decreasing the side effects of prolonged unconjugated hyperbilirubinemia in neonates. It also reduces the duration of phototherapy and thus the duration of stay in the hospital. This research is carried out to improve standard protocol for the management of neonatal hyperbilirubinemia in the local settings.

DETAILED DESCRIPTION:
Complete history and examination will be carried out while patients will be screened for enrollment. After taking informed consent, eligible patients will be selected and divided into two groups A and B by lottery method. Demographics like name, age (hours), gender, birth weight, and gestational age will be noted. Solutions will be prepared in the required strengths and labeled accordingly. Groups A will receive Solution A i.e. Fenofibrate suspension is prepared by dissolving 200 mg capsule in 10 ml distilled water and given as a single dose of 10mg/kg (0.5 ml/kg) and Group B will receive solution B i.e. 0.5ml/ kg normal saline as a placebo. Both groups will receive LED phototherapy under standard conditions. The serum bilirubin level will be noted at the time of admission and then at 12hr, 24hr, and 48 hours of treatment. All this information will be recorded on proforma.

ELIGIBILITY:
INCLUSION CRITERIA:

* Gestational age ≥ 35 weeks
* Birth weight ≥ 2 kg
* Age: 2-7 days of life
* Total serum bilirubin level ≥15mg/dl and ≤20 mg/dl

EXCLUSION CRITERIA:

* Neonates with total bilirubin >20mg/dl
* Conjugated bilirubin level greater than 15% of total serum bilirubin
* Maternal hyperbilirubinemia (on medical record)
* Babies with congenital anomalies (on clinical examination)
* Those not consenting to participate in the study

Ages: 2 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Duration of phototherapy | 6 months
  It is the total time from admission (Serum bilirubin level ≥15 and ≤20 mg/dl) until phototherapy is no longer needed (Serum bilirubin level < 10mg/dl) and is measured in hours.

SECONDARY OUTCOMES:
Serum bilirubin level | 6 months
  It will be measured at the time of admission and then at 12hr, 24hr, and 48 hours of treatment.

IPD SHARING:
Plan to Share IPD: No